CLINICAL TRIAL: NCT05474404
Title: Pilot Study Evaluating the Feasibility of Digitalised Cytolological Slides for Telecytology, Before Implementation in Cameroon
Brief Title: Telecytology as a Triage Tool in LMICs
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: Ecole Polytechnique Fédérale de Lausanne (Other)
Responsible Party: Principal Investigator, Prof. Patrick Petignat, Professor Patrick Petignat, University Hospital, Geneva
Other Study IDs: 2022-00314
Record Dates: First submitted 2022-07-22; First posted 2022-07-26 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Cervical Cancer
Keywords: cytopathology
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cervical smear tests
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cervical smear test — collection of cervical cells using spatula

SUMMARY:
The investigators will collect PAP-test samples from women undergoing colposcopy. Laboratory providers will prepare the samples with a liquid-based cytology method. The providers will then digitalise the slides using a digital scanner. The slides will be sent to cytopathologists who will assess the quality of the slides.

DETAILED DESCRIPTION:
The study will take place over four months. The consultation where the clinician undertakes the colposcopy and takes the additional cytological sample will be the only visit necessary for the patient in relation to the study.

The investigators will require thirty usable cervical samples from the colposcopy clinic of the Maternity of Geneva. The spatula used to take the smear should be immediately transferred to a 10ml sample pot and the head of the spatula should be snapped off and left inside. The investigators will only accept samples that have followed the aformentioned conditions, and it is expected to recruit more than the 30 participants needed if sampling is insufficient. The samples will be prepared by one of 3 laboratory technicians at the same hospital using the manual Surepath® liquid-based preparation method. This includes cell randomization, pipetting and enrichment of diagnostic cervical cells through centrifugation using a settling chamber to create a cellular slide preparation in a circle of 13 mm diameter. The Pap staining procedure is then applied within the chamber.

All thirty glass slides will be scanned and digitalized with a compact portable scanner (Ocus, ®40 by Grundium, Finland). The same laboratory technician who prepared the cervical sample will scan the slide. Ocus ®40 has a 1-slide capacity and permits the acquisition of a whole-slide image as well as robotic microscopy. The scanner features a 12-megapixel image sensor with a 40x objective (numerical aperture: 0.75) and can be connected to a laptop computer over a Wireless Local Area Network (WLAN) connection. To avoid areas being out of focus, the Z-stack modality of acquisition will be used at three focal plane levels with a 1 µ interval. In Europe, Ocus®40 is IVDR certified for diagnostic use.

The ease of the manual preparation method and scanning of slides will be assessed by asking the laboratory technician to rate the difficulty from very easy to very difficult on a 5-point rating scale (score 1= very difficult, 5=very easy) for each preparation step. The time taken for the manual preparation and scanning of glass slides will also be measured with a stopwatch and recorded by the technician.

Quality characteristics of the thirty digitalized slides will be scored as excellent, good, fair, or poor (based on sharpness and visualization through thick cell clusters) by two cytopathologists reading the slides. The time taken to screen digitized slides will be calculated.

In addition, cellularity will be assessed in the preparation area of the glass slide. Under a 40× objective and an eyepiece with a field number of 20, the total number of cells will be computed using the following formula: N=n(acd/amf), where N=total cell count, n=mean cell count of 10 adjacent fields of view along the horizontal diameter in the center of the circle, acd=area of cell deposit and amf=area of microscopic field.

The following data will be recorded and stored for each patient

* the number between 1-30 that has been given to the patient plus previous cytological diagnosis
* the easiness rating for each step of the manual preparation of the slide (lab technician)
* The easiness rating for the scanning/digitalization of the slides (lab technician)
* the quality rating based on sharpness and visualization through thick cell clusters for each slide (cytopathologists)
* the cellularity of each slide (cytopathologists)
* the time taken to prepare (lab technician), digitalize (lab technician) and read (cytopathologists) the slides

There will be a separate form for the laboratory providers and the cytopathologists. The data from the lab technician and the cytopathologists will be subsequently unified.

ELIGIBILITY:
Inclusion Criteria:

* Women aged > 18 who are undergoing colposcopy at the Geneva University Hospitals (HUG)
* Women who are able to give informed consent as documented by signature
* Availability of an adequate sample for analysis

Exclusion Criteria:

* Pregnant women
* Women who have had a hysterectomy
* Women in whom cytology is indicated at time of colposcopy (independently of this study)

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: women aged >18 who are undergoing colposcopy at the Geneva University Hospitals (HUG)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
quality of digitalized slide | 4 months
  Quality of the prepared and digitalised slide as measured by a score allocated by cytopathologists pertaining to sharpness and visualisation through thick cell clusters (scored as excellent (maximal value), good, fair or poor (minimum value)) as well as the cellularity of the slide.

SECONDARY OUTCOMES:
Simplicity of process | 4 months
  - Easiness score allocated by the laboratory providers after the preparation and digitalisation of each slide (1=very difficult; 5=very easy)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No